# Statistical Analysis Plan (SAP)

A Comparison of Tc 99m Tilmanocept Quantitative Imaging with Immunohistochemical (IHC) Analysis of CD206 Expression in Synovial Tissue from Subjects Clinically Diagnosed with Rheumatoid Arthritis (RA)

Study No: NAV3-32

Version 1.0

**September 15, 2022** 

Prepared for Navidea Biopharmaceuticals, Inc. 4995 Bradenton Avenue, Suite 240 Dublin, OH 43017

Prepared by STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 www.statkingclinical.com



## **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

| agree to the format and content of this document. | |
|---|---|
| Michael Rosol, PhD Chief Medical Officer Navidea Biopharmaceuticals 4995 Bradenton Avenue, Suite 240 Dublin, Ohio 43017 MRosol@navidea.com | Oct, 4, 2027 Date |
| Rachael Hershey MS, CCRP Associate Director, Clinical Research & Operatio Navidea Biopharmaceuticals 4995 Bradenton Avenue, Suite 240 | Date Date |

Authored by:

Dublin, Ohio 43017 RHershey@navidea.com

lan Lees, MS Statistician

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 327 ian@statkingclinical.com Approved by (internal review):

Zachary Steckler, MS

Statistician

STATKING Clinical Services

759 Wessel Drive

Fairfield, OH 45014

513-858-2989 ext. 303

zachary@statkingclinical.com

Approved by:

Clare Gerger Clare Geiger, RN **Project Manager** 

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014

513-858-2989 ext. 304

clare@statkingclinical.com

10/4/2022

10.4-2022

# **Revision History**

N/A

# **List of Abbreviations and Definitions of Terms**

| Term | Definition |
|---|---|
| μg | microgram |
| ACR/EULAR | American College of Rheumatology/European League |
| | Against Rheumatism |
| ADR | adverse drug reaction |
| AE | adverse event |
| Anti TNF-α | Anti-Tumor Necrosis Factor $\alpha$ biological Disease Modifying |
| bDMARD | Anti-Rheumatic Drug |
| CDAI | Clinical Disease Activity Index |
| CRF | case report form |
| CSR | clinical study report |
| CT | X-ray computed tomography |
| DAS28 | Disease activity score used with the ACR/EULAR 2010 RA |
| | guidelines |
| ECG | electrocardiogram |
| FDA | Food and Drug Administration |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| HC | healthy controls |
| ICH | International Conference on Harmonization |
| ITA | intent-to-assay |
| IV | intravenous |
| mCi | milliCurie (37x10 <sup>6</sup> becquerels; 37megabecquerels) |
| MCP | metacarpophalangeal |
| MedDRA | Medical Dictionary for Regulatory Activities |
| OA | osteoarthritis |
| PIP | proximal interphalangeal |
| PP | per protocol |
| PT | preferred term |
| RA | rheumatoid arthritis |
| ROI | region of interest |
| RR | reference region |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SOC | system organ class |
| SPECT | single photon emission computed tomography |
| Tc 99m | technetium-99m metastable isotope; γ-emitting (half-life |
| | 6.02 h) |
| tilmanocept | DTPA Mannosyl Dextran (the US Adopted Name for the |
| | drug substance of Lymphoseek) |
| TUV | Tilmanocept uptake value |
| US | United States |

| Term | Definition |
|-----------------|------------------------------------------------------------|
| $\bar{X}_{ROI}$ | the decay-corrected average voxel intensity of a region of |
| | interest |

# **Table of Contents**

| APPROVAL PAGE | 1 |
|------------------------------------------------------|----|
| REVISION HISTORY | 4 |
| LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 5 |
| INTRODUCTION | 9 |
| 1.0 SYNOPSIS OF STUDY DESIGN/PROCEDURES | 9 |
| 1.1 Design and Treatment | 10 |
| 1.2 Study Procedures | 11 |
| 1.3 Sample Size | 12 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 12 |
| 2.1 Types of Analyses | 12 |
| 2.2 Analysis Populations | 12 |
| 2.3 Missing Data Conventions | 13 |
| 2.4 Interim Analyses | 13 |
| 2.6 Study Center Considerations in the Data Analysis | 14 |
| 2.7 Documentation and Other Considerations | 14 |
| 3.0 ANALYSIS OF BASELINE PATIENT CHARACTERISTICS | 15 |
| 4.0 ANALYSIS OF EFFICACY | 15 |
| 4.1 Description of Efficacy Variables | 15 |
| 4.2 Analysis of Efficacy Variables | 16 |
| 5.0 ANALYSIS OF SAFETY | 20 |
| 5.1 Description of Safety Variables | 20 |
| 5.2 Description of Safety Analysis | 20 |

| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 21 |
|---------------------------------------------------------|----|
| 6.1 Patient Completion | 21 |
| 6.3 Study Drug Administration | 22 |
| 6.4 RA Evaluation and Screening Physical Exam | 22 |
| 6.5 Concomitant Medications | 22 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 23 |
| 8.0 REFERENCES | 28 |
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATIONS | 29 |
| APPENDIX R _ TARI F SHELLS | 30 |

#### INTRODUCTION

### Description

This Statistical Analysis Plan (SAP) is consistent with the study protocol Amendment 6 (dated 24 June 2021) and includes the latest details of efficacy and safety summaries to be included in the clinical study report (CSR).

The preparation of this SAP is done in accordance with STATKING Clinical Services SOP SCI 02-54, Statistical Analysis Plans.

# 1.0 Synopsis of Study Design/Procedures

This is a Phase 2b, open-label, multi-center, multinational, non-randomized, single-dose study designed to assess the relationship between quantitative Tc 99m tilmanocept planar imaging and synovial histopathology in subjects clinically diagnosed with RA.

The objectives of the study are:

### **Primary Objectives:**

- Assessment of the relationship between joint-specific tilmanocept uptake value (TUV<sub>joint</sub>) and synovial anatomic pathology.
- IHC assessment of macrophage expression of the CD206 receptor.

#### Secondary Objectives:

- Assessments of CD68 and CD163 receptor expression levels through IHC microscopy.
- Classification of synovial anatomic pathology as
  - Lympho-myeloid
  - Diffuse myeloid
  - Pauci-immune fibroid

#### **Exploratory Objectives:**

- Determine the relationship between TUV<sub>joint</sub> and mRNA expression profiles of CD68, CD163, and CD206 as determined by RNA sequencing (RNA-seq).
- Determine the relationship between TUV<sub>joint</sub> and the number, size, and intensity of CD68, CD163, and CD206 as determined by (optional) flow cytometry.
- Evaluate synovial expression of CD3, CD20, CD55, and TE-7 and CD206 in synovial tissue biopsy specimens.

• Assessment of the relationship between global tilmanocept uptake value (TUV<sub>global</sub>) and synovial anatomic pathology.

#### Safety Objective:

 Evaluate safety through the examination of adverse event (AE) incidence, physical examination findings, and changes over time in laboratory tests, electrocardiograms (ECGs), and vital signs.

#### 1.1 Design and Treatment

Subjects will receive the administration of Tc 99m tilmanocept through an intravenous (IV) route of administration. All subjects will receive a 150  $\mu g$  mass dose of tilmanocept radiolabeled with 10 mCi of Tc 99m and will be at study time 00:00. Following injection, a 10-mL sterile normal saline flush will be administered. The preferred site of IV placement will be the left or right antecubital vein.

Subjects will undergo an imaging assessment of the bilateral hands and wrists followed by an ultrasound-guided synovial biopsy of a select joint at a subsequent visit. Tissue samples from the synovial biopsy procedure will be used for 2 mandatory anatomic pathology evaluations, [1] IHC and [2] RNA-seq, and optional flow cytometry, to provide quantitative and semi-quantitative information regarding joint-specific disease activity. Results from each anatomic pathology evaluation will be correlated with TUV<sub>joint</sub> on planar imaging to mechanistically assess the relationship between synovial anatomic pathology and TUV<sub>joint</sub>.

All joints selected for biopsy will be required to have an ultrasound synovial thickness score of  $\geq 2$ . In instances where more than 1 joint qualifies for biopsy, the candidate joint will be selected based on TUV<sub>joint</sub>.

**Table 1 Biopsy Selection Options** 

| Option | Description |
|--------|--------------------------------------------------|
| 1 | The subject has only 1 |
| | metacarpophalangeal (MCP) joint or |
| | wrist joint with an ultrasound gray- |
| | scale synovitis score of ≥ 2. This joint |
| | will be selected for biopsy. |
| 2 | The subject has 2 or more MCP |
| | and/or wrist joints with an ultrasound |
| | gray-scale synovitis score of ≥ 2. The |
| | joint for biopsy will be selected based |
| | on evaluation of corresponding |
| | TUV <sub>joint</sub> . In the first subject with |
| | multiple qualifying joints, the joint with |

| 46 - 15 1 1 1 - 15 1 1 1 1 1 1 1 1 1 1 1 1 |
|-------------------------------------------------------|
| the highest TUV <sub>joint</sub> will be selected; in |
| the second subject with multiple |
| qualifying joints, the joint with the |
| lowest TUV <sub>joint</sub> will be selected. |
| Selection will proceed in this fashion, |
| alternating between highest and |
| lowest TUV <sub>joint</sub> . |

#### 1.2 Study Procedures

Subjects will be "on study" for up to 45 days depending on the screening window (up to 30 days). The first visit is for the screening (Day -30 to -1). Screening procedures (demographics, vital signs, medical and surgical history, concomitant medications, blood and urine samples for clinical labs, RA specific labs, urine pregnancy testing for subjects of childbearing potential, ultrasound synovitis assessment, AE assessment, and physical exam) will be completed along with RA evaluations including the 2010 ACR/EULAR classification criteria and DAS28 evaluation.

On Day 0 (visit 2) subjects will receive Tc 99m injection and imaging procedures. Pre-injection procedures include the following: Urine pregnancy testing for all women of childbearing potential. Up to 30 minutes prior to study drug administration, an ECG will be performed, followed by assessment of vital signs, AEs, and concomitant medications. After pre-injection procedures are completed, subjects will receive a single IV dose of 150  $\mu g$  of tilmanocept radiolabeled with 10 mCi of Tc 99m. Within 30 minutes after injection, an ECG will be performed, followed by assessment of vital signs and AEs. Between 60 and 75 minutes after injection, subjects will receive an AE assessment and a static gamma camera scan of bilateral hands and wrists. Blood will be drawn for clinical laboratory evaluations after the image acquisition has been completed. Subjects who are administered Tc 99m tilmanocept on Day 0 will be considered to be enrolled in the study.

On the third visit (24-72 hours post-injection), a safety follow-up telephone call will include a review of concomitant medications and an AE check.

On the fourth visit (3-7 days post-injection), subjects will be given an ultrasound assessment of synovitis and then a tissue biopsy of the selected joint in

accordance with Table 1 as described in Section 1.1. In addition, an AE check and a review of concomitant medications will be conducted.

On the fifth and final visit ( $5 \pm 2$  days post-biopsy), a safety follow-up telephone call will include a review of concomitant medications and an AE check.

For the entire study, end of study is defined as last subject last visit.

#### 1.3 Sample Size

The sample size is expected to be approximately 12 to 24 joints. The final sample size will be determined after the completion of an interim analysis including at least 4 subjects in each pathotype (diffuse myeloid, lympho-myeloid and paucimmune fibroid). The final sample size will be chosen based on the sponsor's business requirements regarding precision for the estimated correlation between CD206 expressing macrophage density and  $TUV_{joint}$ . The final sample size will be at least N = 12. If the rarest pathotype has 25% prevalence in the study patient pool, the expected number of subjects at the interim analysis is N = 16. These needs may be further increased because synovial biopsy fails to recover enough tissue for histological analysis in about 15% of cases.

# 2.0 Data Analysis Considerations

## 2.1 Types of Analyses

Data analyses described in this SAP will consist of analyzing efficacy and safety data.

#### 2.2 Analysis Populations

The following analysis populations will be used in the study:

**Safety Population** – The safety population includes all subjects who have been enrolled in the study and injected with Tc 99m tilmanocept regardless of imaging or biopsy status.

**Intent-to-Assay (ITA) Population** – The ITA population includes all subjects that have been enrolled in the study, injected with Tc 99m tilmanocept, received all imaging procedures, and have been biopsied.

**Per-Protocol (PP) Population:** The PP population will include all ITA subjects without major protocol violations. At least 4 evaluable synovial biopsy samples must be available for a subject to be included in the PP population.

## 2.3 Missing Data Conventions

The analysis of the efficacy and safety variables will be carried out on the observed data (i.e., a complete case analysis). For the regression and correlation analyses, a subject must have valid values for all variables to be used in the analysis.

#### 2.4 Interim Analyses

An interim analysis will be performed after 4 subjects in each of the 3 pathotypes (diffuse myeloid, lympho-myeloid, and pauci-immune fibroid) have been imaged. The final sample size will be recalculated after completion of the interim analysis.

#### 2.5 Calculation of TUV

All calculations are done on a reader-specific basis. That is, there is no statistical aggregation of the reader results.

#### **Calculating Joint TUV**

For an individual joint, TUV<sub>joint</sub> is defined as the intrasubject ratio of the average pixel intensity of a joint to the average pixel intensity of the reference region, such that:

$$TUV_{joint} = \frac{\bar{x}_{Joint\ ROI}}{\bar{x}_{PP}}$$

where

- $\bar{X}_{Joint\ ROI}$  is the average pixel intensity of a region of interest (ROI) of a subject at the anterior or posterior view at the time of imaging (nominally 60 minutes);
- $\bar{X}_{RR}$  is the average pixel intensity of the reference region (RR) of a subject at the anterior or posterior view at the time of imaging (nominally 60 minutes).

#### Calculating Global TUV

For each independent blind reader, determine the average TUV<sub>joint</sub> and 95% prediction interval of both the anterior and posterior views of the wrists, MCPs, and PIPs in healthy individuals. For all following calculations, reader specific average TUV<sub>joint</sub> and 95% prediction intervals will be used.

For each RA subject do the following.

Step 1: Calculate TUV<sub>joint</sub> for each of the 22 DAS28 joints for which data are collected.

Step 2: Identify all imaged joints with  $TUV_{joint}$  > upper limit of normal for the anatomically similar joint and view. These will be referred to as inflamed joints (IJ). Each joint has an anterior and posterior view: a joint is considered an IJ if either view has a  $TUV_{joint}$  higher than the upper bound from the normative data set.

Step 3: Calculate the macrophage-involved contribution (MI) to Tc 99m tilmanocept localization for each IJ. This is done by expressing the TUV for the IJ as a fractional change from the mean TUV for the anatomically equivalent joint and view. That is, if TUV<sub>joint</sub> and  $\overline{\mathrm{H}}_{\mathrm{joint}}$  represent the joint and view specific TUV and the mean TUV for the anatomically equivalent joint and view from the normative data set respectively, the macrophage contribution to TUV is MI<sub>joint</sub>:

$$MI_{joint} = \frac{TUV_{joint} - \overline{H}_{joint}}{\overline{H}_{joint}}.$$

Step 4:  $TUV_{global}$  is the total of the macrophage-involved contributions for the IJs. (Note that  $MI_k$  is effectively 0 if  $TUV_{joint}$  is less than or equal to the upper limit of normal from the normative data set.) That is,

$$TUV_{global} = \sum_{All\ IJs} MI_{IJ},$$

$$TUV_{global} = \sum_{k=1}^{22} MI_k.$$

It is presumed that the presence of radiotracer uptake for a joint indicates the presence of activated macrophages. The use of the term "localization" is synonymous with radiotracer uptake.

#### 2.6 Study Center Considerations in the Data Analysis

Up to 10 Centers which include sites in the US, UK, and EU. Analysis will be conducted on the pooled data from all study centers.

#### 2.7 Documentation and Other Considerations

The data analyses described in this SAP will be conducted using SAS<sup>©</sup> Software, version 9.4 or later.

## 3.0 Analysis of Baseline Patient Characteristics

Baseline and demographic characteristics of the safety population will be summarized. Continuous variables (age, height, and weight) will be summarized via mean, standard deviation, minimum, maximum, and number of non-missing responses. Categorical variables (gender, race, and ethnicity) will be summarized via counts and percentages.

A detailed listing of baseline data for each patient in the safety population will also be provided, as shown in Appendix B.

# 4.0 Analysis of Efficacy

## 4.1 Description of Efficacy Variables

## 4.1.1 Primary efficacy variables

The primary efficacy variables for this study are:

- Tc 99m tilmanocept uptake values (TUV<sub>joint</sub>) for the biopsied joints;
- IHC assessment of macrophage expression of the CD206 receptor.

The primary endpoint is:

 The correlation between joint-specific tilmanocept uptake value (TUV<sub>joint</sub>) and the number and area fraction of CD206 expression as determined by IHC assessment.

#### 4.1.2 Secondary efficacy variables

The secondary variables for this study are:

- IHC and immunofluorescence assessment of macrophage expression and co-expression of the CD68 and CD163 receptors.
- Pathotype classification of RA disease as lympho-myeloid, diffuse myeloid, or pauci-immune fibroid, based on TUV<sub>joint</sub>.

The secondary endpoints are:

- The correlation between TUV<sub>joint</sub> and the number and area fraction of CD68 and CD163 determined by IHC assessments.
- Classification of synovial anatomic pathology into Lympho-myeloid, Diffuse myeloid, and Pauci-immune fibroid types as a function of CD68, CD163, CD206, CD3, CD20, CD55, and TE7 expression determined by

IHC assessments using a multinomial logistic regression model with TUV<sub>joint</sub> as a covariate.

The correlation between the expression of CD68, CD163, and CD206.

### 4.1.3 Exploratory efficacy variables

The exploratory variables for this study are:

- IHC assessment of macrophage expression of the CD3, CD20, CD55, and TE7 biomarkers.
- mRNA levels in synovial tissue for the CD206, CD163, and CD68 biomarkers.
- Flow cytometry measurements of CD206, CD163, and CD68 biomarker expression and co-expression.
- Tc 99m tilmanocept global uptake values (TUV<sub>global</sub>) per subject.
- IHC assessment of the expression of a biomarker (e.g., CD206, TE7) is determined from immunofluorescent microscopy, specifically:
  - The ratio of the total fluorescent stained area to the total field area under 4x and 10x power magnification.
- Pathotype classification of RA disease as lympho-myeloid, diffuse myeloid, or pauci-immune fibroid, based on TUV<sub>global</sub>.

The exploratory endpoints for this study are:

- The correlation of the expression of CD3, CD20, CD55, and TE7 with CD206 as measured through IHC.
- The correlation of TUV<sub>joint</sub> with the expression of CD206, CD163, and CD68 as measured through RNA-seq.
- The number and size of CD206, CD163, and CD68 expressing macrophages as measured through (optional) flow cytometry and their correlation with TUV<sub>ioint</sub>.
- The correlation between TUV<sub>global</sub> and synovial anatomic pathology as determined by IHC assessments.
- Classification of synovial anatomic pathology into Lympho-myeloid, Diffuse myeloid, and Pauci-immune fibroid types using a multinomial logistic regression model with TUV<sub>global</sub> as a covariate.

#### 4.2 Analysis of Efficacy Variables

All efficacy analyses will be conducted on both the ITA and PP populations. The ITA population will be the primary analysis set.

## 4.2.1 Primary Efficacy Variables

The primary endpoint will be analyzed by computing the Pearson (product-moment) and Spearman (rank) correlation coefficient between the TUV for the biopsied joint and the final CD206 expressing macrophage count. The CD206 expressing macrophage count is derived from the IHC histopathology and ultrasound imaging:

 The fraction of CD206 expressing macrophages under 4x and 10x power magnification, defined as the ratio of the total fluorescent stained area to total field area. Specifically, area fraction (AF) is defined as

$$AF = \frac{Total\ Stained\ Area}{Total\ Field\ Area} \times 100\%.$$

• The volume of synovial tissue in the biopsied joint, defined as the ultrasound synovial thickness score (Vol). The CD206 macrophage count will be the product of these 2 variables (that is, CD206 = AF\*Vol).

CD206 expressing macrophage fraction and  $TUV_{joint}$  will be summarized with descriptive statistics (number of data pairs, means, standard deviations, minima, medians, and maxima as well as the Pearson correlation between the variables). The ultrasound synovitis score will be summarized with a frequency table. Defining  $\rho$  to be the population correlation coefficient, a test of the hypotheses

$$H_o: \rho \leq 0$$
  
 $H_a: \rho > 0$ 

will be performed using Fisher's Z-transformation and its Normal approximation. A 95% confidence interval for the population correlation coefficient ( $\rho$ ) based on the Fisher Z-transformation (the inverse hyperbolic tangent) and its normal approximation will be provided. The joint distribution of the CD206 macrophage count and TUV<sub>joint</sub> will be summarized graphically with a scatter diagram of the data pairs with the least-squares regression line superimposed on the graph. The joint distribution of the component variables of CD206 macrophage count will be graphically summarized with box plots showing the conditional distribution of TUV<sub>joint</sub> for each category of synovitis score.

## 4.2.2 Secondary Efficacy Variables

Co-expression of the CD68, CD163, and CD206 markers will be analyzed by 2 methods. First, by providing the product-moment and Spearman rank correlation matrices of the IHC field measurements (that is, the fraction of macrophages expressing the markers will not be multiplied by the synovitis score). Descriptive statistics of the data triplets used to calculate the correlation matrices will be

provided (number of data triplets, means, standard deviations, minima, medians, and maxima). In the second method, histological sections will undergo immunofluorescent staining for the 3 markers and DAPI. For each section evaluated, up to 50 cells from the synovial sublining will be identified for each of the 3 markers. For each identified cell (up to 150/section), the rate of coexpression of the 3 markers will be determined. For sections with sparse marker expressing cells, four microscope fields will be randomly selected. Co-expression of the markers will be quantified for any cell observed expressing a marker.

The ability of TUV<sub>joint</sub> to discriminate among lympho-myeloid, diffuse myeloid, and pauci-immune fibroid RA disease types will be evaluated with a multinomial logistic regression model. The model in terms of the logit (log odds) of the outcome is defined as:

$$ln\frac{\pi_j}{1-\pi_j} = \alpha_j + \beta_j X$$

where

j = category of the outcome

 $\frac{\pi_j}{1-\pi_j} = \text{odds}$   $\alpha = \text{intercept}$   $\beta = \text{slope}$ 

 $X = TUV_{joint}$ 

RA type will be the response variable and  $TUV_{joint}$  will be the explanatory variable. ROC curves will be generated using the lympho-myeloid type as the base class. The marginal distribution of disease type will be summarized with a frequency table, while the marginal distribution of  $TUV_{joint}$  will be summarized with descriptive statistics (number of data pairs, mean, standard deviation, minimum, median and maximum). The joint distribution will be graphically summarized with box plots showing the conditional distribution of  $TUV_{joint}$  for each disease type.

### 4.2.3 Exploratory Efficacy Endpoints

Expression of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 biomarkers and their association with TUV<sub>joint</sub> will be assessed with the Pearson (product-moment) and the Spearman (rank) correlation matrices calculated for each measurement of expression (IHC, RNA<sub>seq</sub>, and [optional] flow cytometry). The marginal distributions will be summarized with descriptive statistics (number of complete data points, means, standard deviations, minima, medians, and maxima). The joint distribution will be presented graphically in a windowpane plot of the scatter diagrams.

Expression of CD206, CD163, and CD68 genes in mRNA will be measured with cDNA probes. The TUV<sub>joint</sub> values concentrations will be regressed on the mRNA

abundance as determined by RNA-seq values. The marginal distributions will be summarized with descriptive statistics (number of complete data points, means, standard deviations, minima, medians, and maxima). The joint distribution will be presented with a windowpane plot of the scatter diagrams. The regression coefficients will be presented with the estimated residual covariance matrix. The number, size, and co-expression of CD68, CD163, and CD206 expressing macrophages measured by flow cytometry and their relationship with TUV<sub>joint</sub> will be assessed with the Pearson (product-moment) and Spearman (rank) correlation matrices. The marginal distributions of all variables will be summarized by descriptive statistics (number of complete data points, means, standard deviations, minima, medians, and maxima). The joint distributions will be presented graphically in a windowpane plot of the scatter diagrams.

The ability of TUV<sub>global</sub> to discriminate among lympho-myeloid, diffuse myeloid, and pauci-immune fibroid RA disease types will be evaluated with a multinomial logistic regression model. The model in terms of the logit of the outcome is defined as:

$$ln\frac{\pi_j}{1-\pi_i} = \alpha_j + \beta_j X$$

where

j = category of the outcome

$$\frac{\pi_j}{1-\pi_j}$$
 = odds  
 $\alpha$  = intercept  
 $\beta$  = slope  
 $X$  = TUV<sub>qlobal</sub>

RA type will be the response variable and  $TUV_{global}$  will be the explanatory variable. ROC curves will be generated using the lympho-myeloid type as the base class. The marginal distribution of disease type will be summarized with a frequency table, while the marginal distribution of  $TUV_{global}$  will be summarized with descriptive statistics (number of data pairs, mean, standard deviation, minimum, median and maximum). The joint distribution will be graphically summarized with box plots showing the conditional distribution of  $TUV_{global}$  for each disease type.

If it is found (based on the ROC curves from the multinomial logistic regressions) that  $TUV_{joint}$  and  $TUV_{global}$  can discriminate between the three RA disease types, then no additional analyses will be performed. However, if this is not the case, then two binary logistic regression analyses, with fibroid vs. non-fibroid disease type as the response and  $TUV_{joint}$  and  $TUV_{global}$  as predictors, respectively, will also be conducted.

# 5.0 Analysis of Safety

#### 5.1 Description of Safety Variables

The safety analysis variables are defined as follows:

- Adverse Events (AEs)
- Clinical Laboratory Tests (hematology, serum chemistry, urinalysis)
- ECG Parameters
- Vital Signs

All adverse events (AEs) will be observed for each subject from the time of signing of informed consent until study completion. A treatment-emergent AE (TEAE) is defined as an AE whose start date is on or after the date of the first tilmanocept injection. If the first injection date or the AE start date is missing, the AE will be considered treatment emergent.

Prior to analysis to all AEs will be coded using the MedDRA coding dictionary. Based on the coded terms, TEAEs will be summarized as follows:

- By system organ class (SOC) and preferred term (PT);
- By SOC and PT and relation to the study drug;
- By SOC and PT and severity.

#### 5.2 Description of Safety Analysis

The following describes the safety analyses to be performed for the study. All safety analyses will be performed on the safety population.

Observed and change from baseline for vital sign parameters, ECG parameters, hematology, clinical chemistry, and urinalysis parameters will be summarized using descriptive statistics (n, mean, standard deviation, min, median, and max) at each timepoint.

A data listing will be prepared that reflects the occurrence of TEAEs associated with each concomitant medication or class of medications to examine whether a drug interaction signal is detectable.

## **Clinical Laboratory Tests**

Clinical laboratory tests will be performed at screening and after image acquisition. Abnormal laboratory values will be assessed for clinical significance. For each quantitative laboratory test, descriptive statistics (mean, standard

deviation, median, range, n) on the raw, as well as their changes from baseline, will be presented by timepoint.

If multiple labs were performed at a given visit, then the latest results will be summarized in the analysis tables. All collected lab data will be listed.

#### **ECG Parameters**

A standard 12-lead ECG will be obtained up to 30 minutes before investigational product administration and within 30 minutes after investigational product administration. The ECG will be performed with the subject in a resting position for at least 1 minute. Continuous ECG monitoring is not required. At a minimum, the heart rate, QRS, PR, and QT intervals will be collected. QTc will be calculated using the Fridericia formula.

#### **Vital Signs**

Vital signs will be performed at screening, up to 30 minutes before, and within 30 minutes after investigational product administration. Height and weight will be measured only at screening and will be summarized as part of the baseline and demographic information. For each vital sign (respiration rate, systolic blood pressure, diastolic blood pressure, heart rate, and temperature), descriptive statistics (mean, standard deviation, minimum, maximum, n) on the raw, as well as their changes from baseline, will be presented by timepoint. The baseline value for each of the post-injection vital sign parameters will be the corresponding pre-injection time point. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

# 6.0 Other Relevant Data Analyses/Summaries

#### **6.1 Patient Completion**

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of patients withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The table will include summary counts and percentages. A data listing of all subject completion and withdrawal data will also be constructed.

#### 6.2 Physical Exam

Physical exams will be performed at screening. All physical exam data will be listed.

#### **6.3 Study Drug Administration**

The volume, calculated mass dose, and radioactivity of Tc 99m Tilmanocept injected will be summarized with descriptive statistics. All study drug administration data will be listed.

#### 6.4 RA Evaluation and Screening Physical Exam

Each RA subject will undergo a DAS28 evaluation during screening. The swollen and tender joints will be identified and documented during the physical examination. Results of all DAS28 evaluations will be listed.

#### 6.5 Concomitant Medications

All prior and concomitant medications will be listed, as shown in Appendix B. A separate data listing will be created to show only those medications that were taken for RA within the 6 months prior to Day 0 injection.

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 1 | Subject Disposition | Х | Х |
| 2 | Demographics and Baseline Data Descriptive Statistics - Continuous Variables (Safety Population) | X | X |
| 3 | Demographics and Baseline Data Descriptive Statistics – Categorical Variables (Safety Population) | Х | Х |
| 4 | Descriptive Statistics of TUV <sub>joint</sub> and the CD206<br>Expressing Macrophage Fraction (ITA population) | Х | Х |
| 5 | Descriptive Statistics of TUV <sub>joint</sub> and the CD206<br>Expressing Macrophage Fraction (PP Population) | Х | |
| 6 | Number and Percent of Subject's Ultrasound Synovitis Scores (ITA Population) | X | Х |
| 7 | Number and Percent of Subject's Ultrasound Synovitis Scores (PP Population) | X | |
| 8 | Pearson (Product-Moment) Correlation between CD68, CD163, and CD206 of IHC Measurements (ITA Population) | X | X |
| 9 | Pearson (Product-Moment) Correlation between CD68, CD163, and CD206 of IHC Measurements (PP Population) | X | |
| 10 | Spearman (Rank) Correlation between CD68, CD163, and CD206 of IHC Measurements (ITA Population) | X | |
| 11 | Spearman (Rank) Correlation between CD68, CD163, and CD206 of IHC Measurements (PP Population) | X | |
| 12 | Descriptive Statistics of CD68, CD163, and CD206 from IHC Measurements (ITA Population) | X | X |
| 13 | Descriptive Statistics of CD68, CD163, and CD206 from IHC Measurements (PP population) | X | |
| 14 | Number and Percent of Subjects in Each RA Disease Type - TUV <sub>joint</sub> (ITA Population) | Х | Х |
| 15 | Number and Percent of Subjects in Each RA Disease Type - TUV <sub>joint</sub> (PP Population) | Х | |
| 16 | Number and Percent of Subjects in Each RA Disease<br>Type – TUV <sub>global</sub> (ITA Population) | Х | |
| 17 | Number and Percent of Subjects in Each RA Disease Type – TUV <sub>global</sub> (PP Population) | Х | |
| 18 | Descriptive Statistics of the Marginal Distribution of TUV <sub>joint</sub> (ITA Population) | Х | X |
| 19 | Descriptive Statistics of the Marginal Distribution of TUV <sub>joint</sub> (PP Population) | Х | |
| 20 | Descriptive Statistics of the Marginal Distribution of TUV <sub>global</sub> (ITA Population) | Х | |
| 21 | Descriptive Statistics of the Marginal Distribution of TUV <sub>global</sub> (PP Population) | Х | |
| 22 | Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by IHC Measurement (ITA Population) | X | X |

| Table | Table Title | Included in Final | Shown in Appendix |
|---|---|---|---|
| <b>No.</b> 23 | Table Title Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by IHC Measurement (PP Population) | Tables<br>X | В |
| 24 | Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by RNA <sub>seq</sub> (ITA Population) | X | |
| 25 | Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by RNA <sub>seq</sub> (PP Population) | Х | |
| 26 | Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by Flow Cytometry (ITA Population) | Х | |
| 27 | Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by Flow Cytometry (PP Population) | Х | |
| 28 | Spearman (Rank) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by IHC Measurement (ITA Population) | X | X |
| 29 | Spearman (Rank) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by IHC Measurement (PP Population) | X | |
| 30 | Spearman (Rank) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by RNA <sub>seq</sub> (ITA Population) | Х | |
| 31 | Spearman (Rank) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by RNA <sub>seq</sub> (PP Population) | Х | |
| 32 | Spearman (Rank) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by Flow Cytometry (ITA Population) | Х | |
| 33 | Spearman (Rank) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by Flow Cytometry (PP Population) | Х | |
| 34 | Descriptive Statistics of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> Measured by IHC Measurement (ITA Population) | Х | Х |
| 35 | Descriptive Statistics of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with | Х | |

| Table | | Included in Final | Shown in Appendix |
|---|---|---|---|
| No. | Table Title | Tables | В |
| | TUV <sub>joint</sub> Measured by IHC Measurement (PP Population) | | |
| 36 | Descriptive Statistics of CD3, CD20, CD55, CD68, | Х | |
| | CD163, CD206, and TE7 Biomarkers Association with | , , | |
| | TUV <sub>joint</sub> Measured by RNA <sub>seq</sub> (ITA Population) | | |
| 37 | Descriptive Statistics of CD3, CD20, CD55, CD68, | Х | |
| | CD163, CD206, and TE7 Biomarkers Association with | | |
| | TUV <sub>joint</sub> Measured by RNA <sub>seq</sub> (PP Population) | | |
| 38 | Descriptive Statistics of CD3, CD20, CD55, CD68, | Х | |
| | CD163, CD206, and TE7 Biomarkers Association with | | |
| | TUV <sub>joint</sub> Measured by Flow Cytometry (ITA Population) | | |
| 39 | Descriptive Statistics of CD3, CD20, CD55, CD68, | X | |
| | CD163, CD206, and TE7 Biomarkers Association with | | |
| | TUV <sub>joint</sub> Measured by Flow Cytometry (PP Population) | | |
| 40 | Descriptive Statistics of CD68, CD163, and CD206 | X | X |
| | Genes in mRNA (ITA Population) | | |
| 41 | Descriptive Statistics of CD68, CD163, and CD206 | X | |
| | Genes in mRNA (PP Population) | | |
| 42 | Estimated Residual Covariance with the Regression | X | Х |
| | Coefficients of the CD68, CD163, and CD206 Genes in | | |
| | mRNA (ITA Population) | | |
| 43 | Estimated Residual Covariance with the Regression | Х | |
| | Coefficients of the CD68, CD163, and CD206 Genes in | | |
| | mRNA (PP Population) | | |
| 44 | Pearson (Product-Moment) Correlation of CD68, | X | Х |
| | CD163, CD206 Expressing Macrophages Measured by | | |
| | Flow Cytometry and Their Relationship to TUV <sub>joint</sub> (ITA | | |
| 45 | Population) | | - |
| 45 | Pearson (Product-Moment) Correlation of CD68, | X | |
| | CD163, CD206 Expressing Macrophages Measured by | | |
| | Flow Cytometry and Their Relationship to TUV <sub>joint</sub> (PP | | |
| 46 | Population) Spearman (Rank) Correlation of CD68, CD163, CD206 | Х | |
| 40 | Expressing Macrophages Measured by Flow Cytometry | ^ | |
| | and Their Relationship to TUV <sub>joint</sub> (ITA Population) | | |
| 47 | Spearman (Rank) Correlation of CD68, CD163, CD206 | X | |
| 71 | Expressing Macrophages Measured by Flow Cytometry | _ ^ | |
| | and Their Relationship to TUV <sub>joint</sub> (PP Population) | | |
| 48 | Descriptive Statistics of CD68, CD163, and CD206 | Х | Х |
| 10 | Expressing Macrophages Measured by Flow Cytometry | | |
| | (ITA Population) | | |
| 49 | Descriptive Statistics of CD68, CD163, and CD206 | Х | |
| | Expressing Macrophages Measured by Flow Cytometry | , , | |
| | (PP Population) | | |
| 50 | Descriptive Statistics of TUV <sub>global</sub> by Pathology Type | Х | Х |
| | (ITA Population) | | |
| 51 | Descriptive Statistics of TUV <sub>global</sub> by Pathology Type (PP | Х | |
| - | Population) | | |
| 52 | Vital Signs Descriptive Statistics (Safety Population) | Х | Х |
| 53 | Clinical Laboratory Tests Descriptive Statistics (Safety | Х | Х |
| | Population) | | |

| Table<br>No. | Table Title | Included in Final Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 54 | ECG Parameters Descriptive Statistics (Safety Population) | Х | Х |
| 55 | Summary of Treatment Emergent Adverse Events (Safety Population) | X | X |
| 56 | Number and Percent of Subjects with TEAEs (Safety Population) | X | Х |
| 57 | Descriptive Statistics of TUV <sub>joint</sub> by Fibroid vs. Non-Fibroid Type (ITA Population) | Х | Х |
| 58 | Descriptive Statistics of TUV <sub>joint</sub> by Fibroid vs. Non-Fibroid Type (PP Population) | Х | |
| 59 | Descriptive Statistics of TUV <sub>global</sub> by Fibroid vs. Non-Fibroid Type (ITA Population) | Х | |
| 60 | Descriptive Statistics of TUV <sub>global</sub> by Fibroid vs. Non-Fibroid Type (PP Population) | Х | |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in<br>Appendix<br>B |
|---|---|---|---|
| Fig1 | Scatterplot of the Joint Distribution of CD206 Macrophage Count and TUV <sub>joint</sub> | X | X |
| Fig2 | Boxplots of the Conditional Distribution of TUV <sub>joint</sub> for Each Category of Synovitis Score | X | X |
| Fig3 | Boxplots of the Conditional Distribution of TUV <sub>global</sub> for Each Category of Synovitis Score | X | |
| Fig4 | ROC Curves by RA Disease Type, Logistic Regression with TUV <sub>joint</sub> | Х | Х |
| Fig5 | ROC Curves by RA Disease Type, Logistic Regression with TUV <sub>global</sub> | Х | |
| Fig6 | Conditional Distribution of TUV <sub>joint</sub> by RA Disease Type | Х | Х |
| Fig7 | Joint Distribution of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV <sub>joint</sub> | Х | Х |
| Fig8 | Joint Distribution of CD68, CD163, and CD206 in mRNA | Х | X |
| Fig9 | Joint Distribution of CD68, CD163, and CD206<br>Measured by Flow Cytometry | Х | Х |

| Data<br>Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix<br>B |
|---|---|---|---|
| DL1 | Subject Disposition Data Listing | X | X |
| DL2 | Inclusion/Exclusion Data Listing | Х | X |
| DL3 | Protocol Deviations Data Listing | X | X |
| DL4 | Demographics Data Listing | X | X |
| DL5 | Subjects Excluded from ITA Population Data Listing | X | Х |
| DL6 | Subjects Excluded from PP Population Data Listing | X | X |
| DL7 | Subjects Excluded from Safety Population Data Listing | X | X |
| DL8 | Medical History Data Listing | X | X |
| DL9 | Prior and Concomitant Medications Data Listing | X | X |
| DL10 | Prior and Concomitant RA Medications Data Listing | Х | Х |
| DL11 | Adverse Events Data Listing | X | X |
| DL12 | Occurrence of TEAEs Associated with Concomitant Medications or Class of Medications | Х | Х |
| DL13 | Subject Laboratory Profiles – Hematology Data Listing | Х | Х |
| DL14 | Subject Laboratory Profiles – Serum Chemistry Data<br>Listing | Х | |
| DL15 | Subject Laboratory Profiles – Urinalysis Data Listing | X | |
| DL16 | Subject Laboratory Profiles – Rheumatology Panel Data Listing | Х | |
| DL17 | Physical Exam Data Listing | Х | Х |
| DL18 | ACR/EULAR 2010 Classification Data Listing | Х | Х |
| DL19 | DAS-28 by Joint Data Listing | Х | X |
| DL20 | DAS-28 by Subject Data Listing | Х | Х |
| DL21 | Vital Signs Data Listing | Х | Х |
| DL22 | ECG Parameters Data Listing | Х | Х |
| DL23 | Study Drug Administration Data Listing | Х | Х |
| DL24 | Post-Injection Imaging Data Listing | Х | Х |
| DL25 | TUV Data Listing | Х | Х |
| DL26 | TUV by Pathology Type | Х | Х |
| DL27 | Biomarkers Data Listing | Х | Х |

# 8.0 References

N/A

## **Appendix A – Tables, Figures and Listing Specifications**

#### Orientation

Tables and figures will be displayed in landscape.

#### Margins

Margins will be 1 inch on all sides. Table and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### Headers

The table number will be on the first line of the title. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, 1 line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (DD-MMM-YYYY)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

#### **Table Disclaimer**

The format of the mock tables shown in the appendix of this SAP will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

# Appendix B – Table Shells

Page x of y

Table 1. Subject Disposition
Navidea Biopharmaceuticals - Study No. NAV3-32

| | | 70 | verall |
|-----------------------|-------------------------|----|--------|
| Screen Failures | | | XX |
| Enrolled | | | xx |
| Completed | | XX | (xxx%) |
| Withdrawn | | XX | (xxx%) |
| Reason for Withdrawal | Adverse Event | XX | (xxx%) |
| | Protocol Violation | XX | (xxx%) |
| | Lost to Follow-Up | XX | (xxx%) |
| | Withdrawal of Consent | XX | (xxx%) |
| | Sponsor Discretion | XX | (xxx%) |
| | Investigator Discretion | XX | (xxx%) |
| | Death | XX | (xxx%) |
| | Other | XX | (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 2. Demographics and Baseline Data Descriptive Statistics - Continuous Variables Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

| | Mean | Std Dev | n | Min | Max | Median |
|-----------------|------|---------|-----|-----|-----|--------|
| Age (years) | xxx | xxx | xxx | xxx | xxx | xxx |
| Height (inches) | xxx | xxx | XXX | xxx | xxx | xxx |
| Weight (pounds) | xxx | xxx | xxx | xxx | xxx | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 3. Demographics and Baseline Data Descriptive Statistics - Categorical Variables Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

| Variable | Category | Overall |
|---|---|---|
| Gender | Male<br>Female | xx (xxx%) |
| Race | American Indian or Alaska Native<br>Asian<br>Black or African American<br>Native Hawaiian or Other Pacific Islander<br>White<br>Other | xx (xxx%)<br>xx (xxx%)<br>xx (xxx%)<br>xx (xxx%)<br>xx (xxx%) |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | xx (xxx%)<br>xx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 4. Descriptive Statistics of  $TUV_{joint}$  and the CD206 Expressing Macrophage Fraction Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)

| Measure<br>/Biomarker | Mean | Std<br>Dev | n | Min | Max | Median | Pearson (Product-<br>Moment) Correlation<br>Coefficient | 95% Confidence<br>Limits <sup>a</sup> | Spearman (Rank)<br>Correlation<br>Coefficient | 95% Confidence<br>Limits <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| CD206 | XXX | XXX | XXX | XXX | XXX | xxx | x.xxx | (x.xxx, x.xxx) | x.xxx | (x.xxx, x.xxx) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for the PP Population (Table 5)

<sup>&</sup>lt;sup>a</sup> 95% Confidence limits for the Pearson (Product-Moment) Correlation Coefficient are based on the Fisher Z-Transformation (the inverse hyperbolic tangent) and its normal approximation.

b 95% Confidence limits for the Spearman (Rank) Correlation Coefficient are based on the Fisher Z-Transformation (the inverse hyperbolic tangent) and its normal approximation.

Page x of y

Table 6. Number and Percent of Subject's Ultrasound Synovitis Scores
Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

| Ultrasound | | Number |
|-----------------|-------|--------------|
| Synovitis Score | Visit | (Percentage) |
| 2 | 1 | xxx(xxx%) |
| 2 | 4 | xxx(xxx%) |
| 3 | 1 | xxx(xxx%) |
| 3 | 4 | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for the PP Population (Table 7)

Page x of y

Table 8. Pearson (Product-Moment) Correlation between CD68, CD163, and CD206 of IHC Measurements

Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

Pearson (Product-

| | | Moment) Correlation | 95% Confidence | |
|-------------|-------------|---------------------|----------------|-----|
| Biomarker 1 | Biomarker 2 | Coefficient | Limits | nª |
| CD68 | CD163 | x.xxx | X.XXX | XXX |
| CD163 | CD206 | x.xxx | X.XXX | XXX |
| CD206 | CD68 | x . xxx | x . xxx | xxx |

a Number of data pairs

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table will be repeated for the Spearman (Rank) Correlation Matrix (Table 10). Tables are repeated for the PP Population (Tables 9, 11).
Page x of y

Table 12. Descriptive Statistics of CD68, CD163, and CD206 from IHC Measurements

Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

| Bio | marker | Mean Std Dev | | nª | Min | Max | Median |
|-----|--------|--------------|-----|-----|-----|-----|--------|
| CD6 | 8 | XXX | XXX | xxx | xxx | xxx | xxx |
| CD1 | 63 | xxx | xxx | xxx | xxx | xxx | XXX |
| CD2 | 06 | xxx | xxx | xxx | xxx | xxx | XXX |

Table Format is Repeated for the PP Population (Table 13)

a Number of data triplets
STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 14. Number and Percent of Subjects in Each RA Disease Type -  $TUV_{joint}$  Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)

| | Number (Percent) |
|----------------------|------------------|
| RA Disease Type | of Subjects |
| Lympho-Myeloid | xxx(xxx) |
| Diffuse Myeloid | xxx(xxx) |
| Pauci-immune Fibroid | xxx (xxx) |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Table will be repeated for  $TUV_{qlobal}$  (Table 16). Tables are repeated for the PP Population (Tables 15, 17).

Page x of y

Table 18. Descriptive Statistics of the Marginal Distribution of  $TUV_{joint}$ Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)

| | Mean | Std Dev | nª | Min | Max | Median |
|----------|------|---------|-----|-----|-----|--------|
| TUVjoint | xxx | xxx | XXX | xxx | xxx | xxx |

Source Program: xxxxxxx.sas

Table will be repeated for  $TUV_{global}$  (Table 20). Tables are repeated for the PP Population (Tables 19, 21).

a Number of complete data points STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 22. Pearson (Product-Moment) Correlation of CD3, CD20, CD55, CD68, CD163, CD206, and TE7
Biomarkers Association with TUV<sub>joint</sub> Measured by IHC Measurement
Navidea Biopharmaceuticals - Study No. NAV3-32
ITA Population (N=xxx)

| | Pearson | | |
|---------------------|--------------------------|---------------------|-----|
| Measure | (Product-Moment) | 95% Confidence | |
| /Biomarker | Correlation <sup>a</sup> | Limits <sup>b</sup> | n° |
| ${\tt TUV_{joint}}$ | | | XXX |
| CD3 | X.XXX | (x.xxx, x.xxx) | XXX |
| CD20 | X.XXX | (x.xxx, x.xxx) | XXX |
| XXX | X.XXX | (x.xxx, x.xxx) | XXX |
| about | | ( | |
| CD206 | X.XXX | (x.xxx, x.xxx) | XXX |
| TE7 | x.xxx | (x.xxx, x.xxx) | xxx |
| 111 | A • AAA | (A.AAA, A.AAA) | AAA |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for  $RNA_{seq}$  and Flow Cytometry (Tables 24, 26). Each table will be repeated for the PP Population (Tables 23, 25, 27).

<sup>&</sup>lt;sup>a</sup> Pearson (Product-Moment) correlation between TUV<sub>joint</sub> and the indicated measurement/biomarker.

 $<sup>^{\</sup>mbox{\scriptsize b}}$  Confidence limits calculated using the Fisher Z-transformation.

 $<sup>^{\</sup>mbox{\tiny c}}$  Number of complete data points.

Page x of y

| Measure<br>/Biomarker | Spearman (Rank)<br>Correlation <sup>a</sup> | 95% Confidence<br>Limits <sup>b</sup> | n° |
|---|---|---|---|
| TUVjoint | | | XXX |
| CD3 | x.xxx | (x.xxx, x.xxx) | xxx |
| CD20 | x.xxx | (x.xxx, x.xxx) | xxx |
| xxx | x.xxx | (x.xxx, x.xxx) | xxx |
| CD206 | x.xxx | (x.xxx, x.xxx) | XXX |
| TE7 | x.xxx | (x.xxx, x.xxx) | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for  $RNA_{seq}$  and Flow Cytometry (Tables 30, 32). Each table will be repeated for the PP Population (Tables 29, 31, 33).

<sup>&</sup>lt;sup>a</sup> Spearman (Rank) correlation between TUV<sub>joint</sub> and the indicated measurement/biomarker.

<sup>&</sup>lt;sup>b</sup> Confidence limits calculated using the Fisher Z-transformation.

 $<sup>^{\</sup>mbox{\tiny c}}$  Number of complete data points.

Page x of y

Table 34. Descriptive Statistics of CD3, CD20, CD55, CD68, CD163, CD206, and TE7 Biomarkers Association with TUV<sub>joint</sub> Measured by IHC Measurement

Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

| Measure<br>/Biomarker | nª | Mean | Std Dev | Min | Max | Median |
|-----------------------|-----|------|---------|-----|-----|--------|
| ${ m TUV_{joint}}$ | XXX | xxx | xxx | xxx | xxx | xxx |
| CD3 | xxx | XXX | xxx | XXX | XXX | XXX |
| CD20 | xxx | xxx | xxx | xxx | xxx | XXX |
| xxx | xxx | xxx | xxx | xxx | xxx | xxx |
| CD206 | xxx | xxx | xxx | xxx | xxx | xxx |
| TE7 | XXX | xxx | XXX | xxx | xxx | XXX |

Table Format is Repeated for  $RNA_{seq}$  and Flow Cytometry (Tables 36, 38). Each table will be repeated for the PP Population (Tables 35, 37, 39).

a Number of complete data points.
STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 40. Descriptive Statistics of CD68, CD163, and CD206 Genes in mRNA
Navidea Biopharmaceuticals - Study No. NAV3-32
ITA Population (N=xxx)

| Biomarker | nª | Mean | Std Dev | Min | Max | Median |
|-----------|-----|------|---------|-----|-----|--------|
| CD68 | xxx | xxx | xxx | xxx | xxx | xxx |
| CD163 | xxx | XXX | xxx | XXX | xxx | xxx |
| CD206 | xxx | xxx | xxx | xxx | xxx | xxx |

Table Format is Repeated for the PP Population (Table 41)

a Number of complete data points STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 42. Estimated Residual Covariance with the Regression Coefficients of the CD68, CD163, and CD206

Genes in mRNA

Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

| | Covariance Parameter | Regression |
|-----------------------------------|----------------------|-------------|
| Covariance Parameter <sup>a</sup> | Estimates | Coefficient |
| COV(CD68,CD68) | X.XXX | X.XXX |
| COV(CD163,CD68) | X.XXX | |
| COV(CD163,CD163) | x.xxx | X.XXX |
| COV(CD206,CD68) | x.xxx | |
| COV(CD206,CD163) | x.xxx | |
| COV (CD206, CD206) | x.xxx | x.xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for the PP Population (Table 43)

A least-squares regression model will be implemented with  $TUV_{joint}$  values concentrations as the independent variable and the mRNA abundance as determined by RNA<sub>seq</sub> values as the dependent variables.

a COV = Covariance (i.e. COV(CD163,CD68) = Covariance of CD163 and CD68)

Page x of y

Table 44. Pearson (Product-Moment) Correlation of CD68, CD163, CD206 Expressing Macrophages Measured by Flow Cytometry and Their Relationship to TUVjoint Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

| | Pearson | | | |
|-----------------------|------------------|----------------|-----|---|
| Measure | (Product-Moment) | 95% Confidence | | |
| /Biomarker | Correlationa | Limitsb | n° | - |
| ${ m TUV}_{ m joint}$ | | | XXX | |
| CD68 | x.xxx | (x.xxx, x.xxx) | xxx | |
| CD163 | x.xxx | (x.xxx, x.xxx) | xxx | |
| CD206 | x.xxx | (x.xxx, x.xxx) | xxx | |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for the Spearman (Rank) Correlation Matrix (Table 46). Tables will be repeated for the PP Population (Tables 45, 47).

<sup>&</sup>lt;sup>a</sup> Pearson (Product-Moment) correlation between TUV<sub>joint</sub> and the indicated measurement/biomarker.

b Confidence limits calculated using the Fisher Z-transformation.

<sup>°</sup> Number of complete data points.

Page x of y

Table 48. Descriptive Statistics of CD68, CD163, and CD206 Expressing Macrophages Measured by Flow Cytometry

Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)

| Biomarker | n Mean Std Dev | | Min | Max | Median | Median |
|-----------|----------------|-----|-----|-----|--------|--------|
| CD68 | XXX | xxx | xxx | xxx | xxx | XXX |
| CD163 | xxx | xxx | xxx | xxx | xxx | xxx |
| CD206 | xxx | XXX | xxx | xxx | xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table Format is Repeated for the PP Population (Table 49)

Page x of y

Table 50. Descriptive Statistics of  $TUV_{global}$  by Pathology Type Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)

| Pathology Type | nª | Mean | Std Dev | Min | Max | Median |
|----------------------|-----|------|---------|-----|-----|--------|
| Lympho-myeloid | xxx | xxx | XXX | xxx | xxx | XXX |
| Diffuse myeloid | xxx | XXX | xxx | xxx | xxx | xxx |
| Pauci-immune fibroid | XXX | XXX | XXX | xxx | xxx | XXX |

Table Format is Repeated for the PP Population (Table 51)

a Number of complete data points STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Table 52. Vital Signs Descriptive Statistics
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Vital Sign Parameter | Data | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|
| (units) | Visit | Typea | n | Dev | Mean | Min | Max | Median |
| xxxxxxxxxxxxxxx (xxx) | Screening | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Pre Admin | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Post Admin | Raw | XXX | XXX | xxx | XXX | XXX | XXX |
| | | CFB | XXX | XXX | xxx | XXX | XXX | XXX |
| xxxxxxxxxxxxxxx (xxx) | Screening | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Pre Admin | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Post Admin | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| xxxxxxxxxxxxxxx (xxx) | Screening | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Pre Admin | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Post Admin | Raw | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

<sup>&</sup>lt;sup>a</sup> RAW = data recorded in database; CFB = change from baseline = (parameter value at the current time point)-(Baseline parameter value). STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxxx.sas

| | | Data | | Std | | | | |
|---|---|---|---|---|---|---|---|---|
| Laboratory Test | Visit | Typeª | n | Dev | Mean | Min | Max | Median |
| XXXXXXXXXXXXXXXX | Screening | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 0 - 60 to 75 Minutes Post Admin | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| xxxxxxxxxxxxxxx | Screening | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 0 - 60 to 75 Minutes Post Admin | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| xxxxxxxxxxxxxx | Screening | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | Day 0 - 60 to 75 Minutes Post Admin | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

a RAW = data recorded in database; CFB = change from baseline = (parameter value at the current time point)-(Baseline parameter value).

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table 54. ECG Parameters Descriptive Statistics
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| | | Data | | Std | | | | |
|---|---|---|---|---|---|---|---|---|
| ECG Parameter (units) | Visit | Typeª | n | Dev | Mean | Min | Max | Median |
| xxxxxxxxxxxxxxx (xxx) | Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | 30 Minute Post Admin | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

<sup>&</sup>lt;sup>a</sup> RAW = data recorded in database; CFB = change from baseline = (parameter value at the current time point)-(Baseline parameter value). STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 55. Summary of Treatment Emergent Adverse Events
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| | Overall |
|---|---|
| Subjects with at Least One Treatment Emergent Adverse Event (TEAE) | xxx (xxx%) |
| Maximum TEAE Severity Grade | |
| Mild | xxx (xxx%) |
| Moderate | xxx (xxx%) |
| Severe | xxx (xxx%) |
| <pre>Highest Relationship of TEAE to Study Drug Definitely Not [n(%)] Probably Not [n(%)] Possibly [n(%)] Probably [n(%)] Definitely [n(%)]</pre> | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |
| Highest Relationship of TEAE to Study Procedure | |
| Definitely Not [n(%)] | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Table 56. Number and Percent of Subjects with TEAEs
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Adverse Event Categorya: | Overall |
|---|---|
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%) xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxxx.sas

Table 57. Descriptive Statistics of  $TUV_{joint}$  by Fibroid vs. Non-Fibroid Type Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)

| Type | n <sup>a</sup> | Mean | Std Dev | Min | Max | Median |
|-------------|----------------|------|---------|-----|-----|--------|
| Fibroid | xxx | xxx | xxx | xxx | xxx | xxx |
| non-Fibroid | xxx | xxx | xxx | xxx | xxx | xxx |

Table Format is Repeated for  $TUV_{global}$  (Table 59). Tables will be repeated for the PP Population (Tables 58, 60).

a Number of complete data points STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Figure 1. Scatterplot of the Joint Distribution of CD206 Macrophage Count and TUVjoint Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Figure 2. Boxplots of the Conditional Distribution of  $TUV_{joint}$  by Synovitis Score Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Table Format is Repeated for  $\mathtt{TUV}_{\mathtt{global}}$  (Figure 3).

Page x of y

Figure 4. ROC Curves by RA Disease Type, Logistic Regression with  $TUV_{\text{joint}}$  Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Table Format is Repeated for  $\text{TUV}_{\text{global}}$  (Figure 5).

Page x of y

Figure 6. Conditional Distribution of  $TUV_{joint}$  by RA Disease Type Navidea Biopharmaceuticals - Study No. NAV3-32 ITA Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY)

Page x of y



STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Figure 8. Joint Distribution of CD68, CD163, and CD206 in mRNA
Navidea Biopharmaceuticals - Study No. NAV3-32
ITA Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Figure 9. Joint Distribution of CD68, CD163, and CD206 Measured by Flow Cytometry

Navidea Biopharmaceuticals - Study No. NAV3-32

ITA Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 1. Subject Disposition Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32

| Subject<br>No. | Disposition Status | Date of<br>Completion/<br>Withdrawal/Screen<br>Fail | Withdrawal Reason |
|---|---|---|---|
| xxxx | xxxxxxxxxxxxxxxxxx | xxxxxxxx | ******** |
| XXXX | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 2. Inclusion/Exclusion Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32

| Subject<br>No. | Did Subject<br>Meet All<br>Eligibility<br>Criteria? | Criterion Category | Criterion | Was a<br>Waiver<br>Granted? | Is Subject a<br>Screen<br>Failure? |
|---|---|---|---|---|---|
| XXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |
| XXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx | xxxxxxxx | XXXX | xxxx |
| XXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| XXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 3. Protocol Deviations Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32

| Subject<br>No. | Date of<br>Deviation | Deviation Description | Deviation Category<br>(Major/Minor) |
|---|---|---|---|
| xxxx | xxxxxx | ****** | xxxxxxxxx |
| xxxx | xxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX |
| XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX |
| XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 4. Demographics Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Subject<br>No. | Informed<br>Consent<br>Date/Time | Date<br>of<br>Birth | Height<br>(inches) | Weight<br>(pounds) | Age<br>(yrs) | Gender | Race | Ethnicity |
|---|---|---|---|---|---|---|---|---|
| XXXX | XXXXXX | XXXXXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 5. Subjects Excluded from ITA Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
All Enrolled Subjects (N=xxx)

| Subject No. | Reason for Exclusion |
|-------------|-----------------------------|
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| xxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 6. Subjects Excluded from PP Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
All Enrolled Subjects (N=xxx)

| Subject No. | Reason for Exclusion |
|-------------|-----------------------------|
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| xxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 7. Subjects Excluded from Safety Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
All Enrolled Subjects (N=xxx)

| Subject No. | Reason for Exclusion |
|-------------|-----------------------------|
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| xxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 8. Medical History Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

| | MedDRA System Organ Classa/ | | | |
|---|---|---|---|---|
| Subject | MedDRA Preferred Term/ | | Resolution/Stop | |
| No. | CRF Verbatim Term | Start Date | Date | Ongoing? |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | xxxxxx | XXX |

<sup>&</sup>lt;sup>a</sup> Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

## Data Listing 9. Prior and Concomitant Medications Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

Drug Preferred Terma/ Verbatim/

| | VELDACINI/ | | | | | | |
|---|---|---|---|---|---|---|---|
| Subject | ATC Level 1 Text/ | | | Start | Stop | | |
| No. | ATC Level 4 Text | Indication | Frequency | Date | Date | Route | Ongoing? |
| | | | | | | | _ |
| XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |

<sup>&</sup>lt;sup>a</sup> Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 10. Prior and Concomitant RA Medications Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

Drug Preferred Term<sup>a</sup>/ Verbatim/ Indication/

| | Indication/ | | | | | |
|---|---|---|---|---|---|---|
| Subject | ATC Level 1 Text/ | | Start | Stop | | |
| No. | ATC Level 4 Text | Frequency | Date | Date | Route | Ongoing? |
| • | | | | | | |
| XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
| XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |

<sup>&</sup>lt;sup>a</sup> Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 11. Adverse Events Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| | | Start Date | | | | | |
|---|---|---|---|---|---|---|---|
| | Start | and Time of | MedDRA System | | | | |
| | Date and | Nearest | Organ Class <sup>a</sup> / | | Relation to | | |
| | Time/ | Previous | MedDRA Preferred | | Tc-99m | | |
| Subject | End Date | tilmanocept | Term/ | | tilmanocept/ | | |
| No. | and Time | Injection | CRF Verbatim Term | Severity | Procedure | Serious? | Outcome |
| XXXXXXXX | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxxx | XXXXXXX | xxxxxxxx/ | XXX | XXXXXXXX |
| | xxxxxxx/ | XXXXXXX | xxxxxxxxxxxxxxx | | XXXXXXXX | | |
| | XXXXXXX | | xxxxxxxxxxxxxxx | | | | |
| | XXXXXXX | | | | | | |
| XXXXXXXX | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxxx | XXXXXXXX | xxxxxxxx/ | XXX | XXXXXXXX |
| | xxxxxxx/ | XXXXXXX | xxxxxxxxxxxxxxx | | XXXXXXXX | | |
| | XXXXXXX | | xxxxxxxxxxxxxxx | | | | |
| | XXXXXXX | | | | | | |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 12. Occurrence of TEAEs Associated with Concomitant Medication or Class of Medications

Data Listing

Navidea Biopharmaceuticals - Study No. NAV3-32

Safety Population (N=xxx)

| | | Start Date | | |
|---|---|---|---|---|
| | Start | and Time of | MedDRA System | |
| | Date and | Nearest | Organ Class <sup>a</sup> / | |
| | Time/ | Previous | MedDRA Preferred | Concomitant Medication or |
| Subject | End Date | tilmanocept | Term/ | Class of Medications |
| No. | and Time | Injection | CRF Verbatim Term | Associated with AE |
| XXXXXXXX | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxx | XXXXXXX |
| | xxxxxxx/ | XXXXXXX | xxxxxxxxxxxxxx | |
| | XXXXXXX | | xxxxxxxxxxxxxxx | |
| | xxxxxx | | | |
| xxxxxxxx | xxxxxxx | xxxxxxx | ****** | xxxxxxx |
| | xxxxxxx/ | xxxxxxx | xxxxxxxxxxxxxxx | |
| | xxxxxxx | | xxxxxxxxxxxxxxx | |
| | xxxxxxx | | | |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas
Page x of y

Data Listing 13. Subject Laboratory Profiles - Hematology Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| | | | | | Normal | l Range | |
|---|---|---|---|---|---|---|---|
| Subject | 771 - 11 | Sample Date | Tab Danamakan (Haliba) | D 1 - | T - 1- T | Tab III'ab | |
| No. | Visit | and Time | Lab Parameter (Units) | Result | Lab Low | Lab High | Clin. Sig? |
| XXXX | XXXXXXX | xxxxxxxx / xx:xx | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format is repeated for Serum Chemistry, Urinalysis, and Rheumatology Panel Listings (Listings 14, 15, 16).

Page x of y

Data Listing 17. Physical Exam Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Subject | | Date | | | |
|---|---|---|---|---|---|
| No. | Visit | Conducted | Body System | Result | Abnormality |
| XXXX | XXXXXXX | XXXXXXX | General Appearance | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Skin | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Eyes, Ears, Nose, Throat | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Head and Neck | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Lungs | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Heart | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Abdomen | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Lymph Nodes | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Musculoskeletal | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Nervous System | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | Other: XXXXXX | xxxxxxx | ******* |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 18. ACR/EULAR 2010 Classification Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

### ACR/EULAR 2010

| Subject<br>No. | Visit | Date | Joint<br>Involvement | Serology | Acute-<br>Phase<br>Reactants | Duration<br>of<br>Symptoms | Total Score |
|---|---|---|---|---|---|---|---|
| xxxx | xxxxxxx | xxxxxxx | xxx | xxx | xxx | xxx | xxx |
| xxxx | xxxxxx | xxxxxxx | xxx | XXX | xxx | xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 19. DAS-28 By Joint Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

### DAS28 Joint Classification

| Subject | | | | Result | Result |
|---------|---------|---------|----------|--------------|-------------|
| No. | Visit | Date | Joint | (Right Body) | (Left Body) |
| XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 20. DAS-28 By Subject Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| | | | | | DAS28 | | |
|---|---|---|---|---|---|---|---|
| | | • | | | Patient | | |
| | | | Tender | Swollen | VAS | C-reactive | |
| Subject | | | Joint | Joint | Global | Protein (CRP; | DAS28 |
| No. | Visit | Date | Count | Count | (mm) | mg/L) | Score |
| xxxx | xxxxxx | xxxxxx | xxx | xxx | xxx | xxx | XXX |
| XXXX | xxxxxx | XXXXXX | XXX | xxx | XXX | xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 21. Vital Signs Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Subject<br>No. | Visit | Date | Time | Temp. | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Heart<br>Rate<br>(bpm) | Respirations<br>per Minute |
|---|---|---|---|---|---|---|---|---|
| xxxx | xxxxxx | xxxxxx | xxxxx | xxx | XXX | xxx | xxx | xxx |
| xxxx | xxxxxx | xxxxxx | **** | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx |
| | | | xxxxx | xxx<br>xxx | XXX | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 22. ECG Parameters Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| verall<br>pretation | | QTcF<br>Interval | OT Interval | QRS<br>Interval | PR Interval | Heart Rate | Time | Date | Visit | Subject<br>No. |
|---|---|---|---|---|---|---|---|---|---|---|
| Р | Incerp | Interval | Q'l' Interval | Interval | rk ilitervar | neart Rate | TIME | Date | VISIC | No. |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 23. Study Drug Administration Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Subject<br>No. | Date/<br>Time of<br>Injection | Anatomic<br>Location<br>of<br>Injection | Pre-Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Post-<br>Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Calculated Amount of Administered Radioactivity (mCi) | Calculated<br>Mass Dose<br>(µg) | Volume<br>Injected<br>(mL) | Lot<br>Number |
|---|---|---|---|---|---|---|---|---|
| | / | | / | / | | | | |
| XXXX | xxxxxxxx/<br>xxxx | XXXXXXX | xxx/<br>xxxx | xxx/<br>xxxx | XXX | XXX | XXX | XXX |
| | , | | , | , | | | | |
| XXXX | xxxxxxx/ | XXXXXXXX | xxx/ | xxx/ | XXX | XXX | XXX | XXX |
| | XXXX | | XXXX | XXXX | | | | |
| | xxxxxxxx/ | xxxxxxx | xxx/ | xxx/ | xxx | xxx | XXX | xxx |
| | xxxx | | xxxx | xxxx | | | | |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 24. Post-Injection Imaging Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-32
Safety Population (N=xxx)

| Subject<br>No. | Visit | Date of<br>Imaging | Start Time of Imaging | Planar Imaging<br>Performed? |
|---|---|---|---|---|
| xxxx | xxxxxxx | xxxxxx | xx:xx | XXX |
| xxxx | xxxxxxx | xxxxx | xx:xx | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

# Data Listing 25. TUV Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

| Subject<br>No. | Visit | Date / Time | Region of<br>Interest <sup>a</sup> | TUV | Upper Limit of<br>Normal | Mean of<br>Normal |
|---|---|---|---|---|---|---|
| xxxx | xxxxxx | xxxxxxx / xx:xx | xxxxxx | xxxxx | XXX | xxx |
| xxxx | xxxxxxx | xxxxxxx / xx:xx | xxxxxx | xxxxx | xxx | xxx |

<sup>&</sup>lt;sup>a</sup> Region of Interest is joint or global. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

### Data Listing 26. TUV<sub>global</sub> by Pathology Type Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

| Subject<br>No. | Visit | Date / Time | Pathology Type | $\mathrm{TUV}_{\mathtt{global}}$ | Upper Limit of<br>Normal | Mean of<br>Normal |
|---|---|---|---|---|---|---|
| xxxx | xxxxxx | xxxxxxxx / xx:xx | xxxxx | xxxxx | XXX | xxx |
| xxxx | xxxxxxx | xxxxxxxx / xx:xx | xxxxxx | xxxxx | xxx | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

# Data Listing 27. Biomarkers Data Listing Navidea Biopharmaceuticals - Study No. NAV3-32 Safety Population (N=xxx)

| Subject | | | | Anatomic Pathology | |
|---|---|---|---|---|---|
| No. | Visit | Date / Time | Biomarker | Evaluation | Result |
| xxxx | xxxxxxx | xxxxxxx / xx:xx | xxxxx | xxxx | xxxxx |
| xxxx | xxxxxxx | xxxxxxxx / xx:xx | xxxxx | xxxxx | xxxxx |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas